CLINICAL TRIAL: NCT02824640
Title: Patient-Centered Models of HCV Care for People Who Inject Drugs
Acronym: HERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Massachusetts General Hospital (Other); University of Rhode Island (Other); Johns Hopkins University (Other); West Virginia University (Other); University of New Mexico (Other); University of California (Other); University of Washington (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5723
Record Dates: First submitted 2016-06-23; First posted 2016-07-07 (Estimated); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis C; Medication Adherence
Keywords: Addiction; Adherence; Adverse Effects; Direct Acting Antiviral Agent; Chronic Hepatitis C; Resistance Development; Methadone Clinic; Primary Care; Directly Observed Therapy; Randomized Controlled Trial; Resistance; Reinfection; Treatment Outcome; Patient Navigation; Multi-Site; Liver Disease; Intervention; Sustained Viral Response
MeSH Terms: conditions — Hepatitis C; Medication Adherence; Behavior, Addictive; Hepatitis C, Chronic; Directly Observed Therapy; Reinfection; Liver Diseases | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (Active Comparator): The study will follow a PN model (Check Hep C) developed by NYCDOH in collaboration with Montefiore and the community. HCV PNs will provide the following interventions to those randomized to the PN arm: coordination of HCV treatment; health promotion; assisting patients to overcome barriers; and psychosocial support.
  Health Promotion Sessions: PNs will deliver 4 standardized health promotion sessions to all patients either individually or within a group.
  Optional Weekly Support Groups: Subjects randomized to the PN arm will be offered weekly support groups led by Peers.
  Interventions: Behavioral: Patient Navigation
- modified Directly Observed Therapy (Active Comparator): OAT clinic setting: Observation of HCV medications will be linked to methadone visits among patients receiving methadone. Patients will be receiving methadone as part of routine clinical care for opioid addiction and not as an intervention related to this study. The schedule of five days per week will be considered modified DOT (mDOT). Subjects will initiate HCV treatment on Mondays if feasible. Take home medications will be packed in a weekly electronic blister pack.
  Community health clinic setting: This intervention is considered modified DOT (mDOT) since between 3-5 weekly doses will be directly observed. A minimum of one dose will be observed in person by clinic/study staff. For the remaining observed doses, the research staff and provider will present the participant with a menu of options and determine what will work best for that participant.
  Interventions: Behavioral: modified Directly Observed Therapy

INTERVENTIONS:
Behavioral: Patient Navigation — The study will follow a PN model (Check Hep C) developed by NYCDOH in collaboration with Montefiore and the community. HCV PNs will provide the following interventions to those randomized to the PN arm: coordination of HCV treatment; health promotion; assisting patients to overcome barriers; and psychosocial support.
  Other Names: PN
  Arms: Patient Navigation
Behavioral: modified Directly Observed Therapy — Subjects will be observed taking medications, a minimum of 5 times a week for those enrolled in the OAT setting, and a minimum of 3 times a week for those enrolled in the community health clinic setting.
  Other Names: mDOT
  Arms: modified Directly Observed Therapy

SUMMARY:
People who inject drugs (PWID) have higher rates of hepatitis C virus (HCV) than do other groups. Effective, safe new treatments called direct-acting antiviral agents (DAAs) have been developed recently. Unfortunately, PWID rarely get these treatments. The drugs are expensive, so insurers often do not cover the cost of DAAs. Sometimes providers hesitate to prescribe DAAs because they are concerned that PWID won't take their medication or that these patients might become reinfected.

Several good models for treating PWID exist. One of them is to provide directly observed treatment (DOT). Another model provides treatment to PWID with the support of patient navigators (PN), public health workers who offer support and education to patients. Though both the DOT and PN models have been successful, we still don't know which model works best.

In this study, the investigators will study both DOT and PN models for treating HCV in PWID. The investigators' goal is to find out which model produces the best results and is preferred by patients. Up to 1,000 HCV-infected PWID will participate in the study in eight sites around the country. Patients will be randomized into either the PN or the DOT groups. Patients who end up in the PN group will get a biweekly blister pack of medication to take home. Their PN will provide education and support. The investigators will find out whether patients adhered to medication using an electronic adherence monitoring system. Patients who are randomly assigned to the DOT group will take their medication in front of a staff member.

DETAILED DESCRIPTION:
This is a multi-site national study (8 U.S. cities), where up to 1000 HCV-infected PWIDs (injecting illicit substances within the last 3 months) will be randomized to either PN plus biweekly blister pack dispensation versus mDOT. Among patients who go on to initiate HCV treatment (n=600 targeted) with a once-daily combination regimen, a comparison will be conducted of the proportion of patients in each arm who: (a) optimally adhere (>=80%), (b) complete treatment, (c) achieve SVR, and (d) develop resistance. The primary outcome will be SVR. The 8 sites offer geographic and policy diversity: New York City, Baltimore, Providence, Boston, Morgantown, Seattle, San Francisco, and Albuquerque.

Participants will be recruited from diverse venues: OAT clinics, community health centers, syringe exchange programs, community-based organizations, homeless programs, and cohorts established by research studies. The clinical sites will determine eligibility based on clinical records, or on-site testing including for HCV tests (anti-HCV and HCV viremia) and drug toxicology testing as needed. Study participants will be screened, consented and enrolled on-site at OAT and non-OAT clinic settings.

Patients will be randomized to one of two models of care: patient navigation (PN) vs. modified directly observed treatment (mDOT). Patients enrolled from OAT clinics who are receiving methadone and randomized to mDOT will receive doses of once daily medication at the same time as they receive methadone. Patients enrolled from community health settings and randomized to mDOT may receive observed doses in a range of settings including: at their clinic, at home, a community site (e.g. at a coffee shop or other gathering place), or using a mobile health app on a smartphone. Subjects randomized to PN will receive a standardized PN intervention and additional support through a peer-led support group.

Participants will be followed for up to 140 weeks: 12 weeks of pre-treatment evaluation, 12 weeks of treatment, 12 weeks of follow-up to determine SVR12, and 104 weeks of follow-up to determine long-term SVR and reinfection. Data sources will include clinical lab and imaging results from medical records, blood tests (HCV viral load during long-term follow-up and resistance assays), urine toxicology, questionnaires, electronic monitors for assessing adherence, and interview.

ELIGIBILITY:
Inclusion Criteria:

* HCV infection
* Actively injecting drugs (any substance within 3 months)
* Not previously treated with HCV direct-acting antiviral medications
* Age 18 - 70
* Willing to receive HCV treatment with sofosbuvir/velpatasvir
* Willing to be randomized to either PN vs mDOT
* If receiving methadone, be attending methadone clinic a minimum of 5 times per week
* Able to provide informed consent
* English or Spanish fluency

Exclusion Criteria:

* Pregnant or breast feeding
* Hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Litwin, MD, MPH, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Alain Litwin, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pericot-Valverde I, Lopes SS, Obeysekare J, Batchelder AW, Groome M, Taylor LE, Page K, Tsui JI, Lum PJ, Mehta SH, Feinberg J, Kim AY, Norton BL, Arnsten J, Baker A, Heo M, Litwin AH; HERO Study Group. Depression profiles and hepatitis C treatment outcomes among people who inject drugs: The HERO study. J Psychosom Res. 2025 Dec;199:112417. doi: 10.1016/j.jpsychores.2025.112417. Epub 2025 Oct 17. PMID 41124945
- [Derived] Tsui JI, Ludwig-Barron NT, James JR, Heo M, Sivaraj LB, Arnsten J, Lum PJ, Taylor LE, Mehta SH, Falade-Nwulia O, Feinberg J, Kim AY, Norton B, Page K, Litwin AH. Current Self-reported Pain Before and After Cure of Hepatitis C Among Persons Who Actively Inject Drugs. J Addict Med. 2025 May-Jun 01;19(3):248-253. doi: 10.1097/ADM.0000000000001398. Epub 2024 Oct 30. PMID 39475112
- [Derived] Litwin AH, Tsui JI, Heo M, Mehta SH, Taylor LE, Lum PJ, Feinberg J, Kim AY, Norton BL, Pericot-Valverde I, Arnsten J, Meissner P, Karasz A, McKee MD, Ward JW, Johnson N, Agyemang L, Stein ES, Thomas A, Borsuk C, Blalock KL, Wilkinson S, Wagner K, Carty J, Murray-Krezan C, Anderson J, Jacobsohn V, Luetkemeyer AF, Falade-Nwulia O, Groome M, Davies S, Costello K, Page K; HERO Study Group. Hepatitis C Virus Reinfection Among People Who Inject Drugs: Long-Term Follow-Up of the HERO Study. JAMA Netw Open. 2024 Aug 1;7(8):e2430024. doi: 10.1001/jamanetworkopen.2024.30024. PMID 39186268
- [Derived] Heo M, Norton BL, Pericot-Valverde I, Mehta SH, Tsui JI, Taylor LE, Lum PJ, Feinberg J, Kim AY, Arnsten JH, Sprecht-Walsh S, Page K, Murray-Krezan C, Anderson J, Litwin AH; HERO Study Group. Optimal hepatitis C treatment adherence patterns and sustained virologic response among people who inject drugs: The HERO study. J Hepatol. 2024 May;80(5):702-713. doi: 10.1016/j.jhep.2023.12.020. Epub 2024 Jan 17. PMID 38242324
- [Derived] Tsui JI, Lum PJ, Taylor LE, Mehta SH, Feinberg J, Kim AY, Norton BL, Niu J, Heo M, Arnsten J, Pericot-Valverde I, Thomas A, Blalock KL, Radick A, Murray-Krezan C, Page K, Litwin AH; HERO Study Group. Injecting practices during and after hepatitis C treatment and associations with not achieving cure among persons who inject drugs. Drug Alcohol Depend. 2023 Jun 1;247:109878. doi: 10.1016/j.drugalcdep.2023.109878. Epub 2023 Apr 17. PMID 37150144
- [Derived] Litwin AH, Lum PJ, Taylor LE, Mehta SH, Tsui JI, Feinberg J, Kim AY, Norton BL, Heo M, Arnsten J, Meissner P, Karasz A, Mckee MD, Ward JW, Johnson N, Pericot-Valverde I, Agyemang L, Stein ES, Thomas A, Borsuk C, Blalock KL, Wilkinson S, Wagner K, Roche J, Murray-Krezan C, Anderson J, Jacobsohn V, Luetkemeyer AF, Falade-Nwulia O, Page K; HERO Study Group. Patient-centred models of hepatitis C treatment for people who inject drugs: a multicentre, pragmatic randomised trial. Lancet Gastroenterol Hepatol. 2022 Dec;7(12):1112-1127. doi: 10.1016/S2468-1253(22)00275-8. PMID 36370741

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Navigation: The study will follow a PN model (Check Hep C) developed by NYCDOH in collaboration with Montefiore and the community. HCV PNs will provide the following interventions to those randomized to the PN arm: coordination of HCV treatment; health promotion; assisting patients to overcome barriers; and psychosocial support.
  Health Promotion Sessions: PNs will deliver 4 standardized health promotion sessions to all patients either individually or within a group.
  Optional Weekly Support Groups: Subjects randomized to the PN arm will be offered weekly support groups led by Peers.
  Patient Navigation: The study will follow a PN model (Check Hep C) developed by NYCDOH in collaboration with Montefiore and the community. HCV PNs will provide the following interventions to those randomized to the PN arm: coordination of HCV treatment; health promotion; assisting patients to overcome barriers; and psychosocial support.
- Modified Directly Observed Therapy: OAT clinic setting: Observation of HCV medications will be linked to methadone visits among patients receiving methadone. Patients will be receiving methadone as part of routine clinical care for opioid addiction and not as an intervention related to this study. The schedule of five days per week will be considered modified DOT (mDOT). Subjects will initiate HCV treatment on Mondays if feasible. Take home medications will be packed in a weekly electronic blister pack.
  Community health clinic setting: This intervention is considered modified DOT (mDOT) since between 3-5 weekly doses will be directly observed. A minimum of one dose will be observed in person by clinic/study staff. For the remaining observed doses, the research staff and provider will present the participant with a menu of options and determine what will work best for that participant.
  modified Directly Observed Therapy: Subjects will be observed taking medications, a minimum of 5 times a week for those enrolled in the OAT setting, and a minimum of 3 times a week for those enrolled in the community health clinic setting.
Period: Overall Study
Arm/Group | Patient Navigation | Modified Directly Observed Therapy
Started | 379 | 376
Completed | 264 | 251
Not Completed | 115 | 125

BASELINE CHARACTERISTICS:
Population: mITT, modified intention-to-treat population, which included participants who were randomly assigned and initiated treatment;
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigation | Modified Directly Observed Therapy | Total
Number analyzed (Participants) | 379 | 376 | 755
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 43.1 [34.1 to 51.0] | 43.6 [34.4 to 53.7] | 43.4 [34.2 to 52.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 109 | 218
  Male | 270 | 267 | 537
Race/Ethnicity, Customized [Number; unit: race]
  White/Caucasian | 250 | 226 | 476
  Black/African American | 37 | 66 | 103
  Other | 81 | 70 | 151
  Missing | 11 | 14 | 25
Urine Drug Screen Results at Baseline [Number; unit: urine drug tests]
  Positive for Any drug | 329 | 326 | 655
  Negative for Any Drug | 15 | 12 | 27
  Missing | 35 | 38 | 73

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response (SVR)
Description: HCV viral load undetectable 12 weeks after treatment completion.
Time Frame: 12 weeks after treatment completion
Population: The total N=755 is the number of participants who was randomized between modified Directly Observed Therapy (mDOT) and Patient Navigation (PN) study arms. This sample is referred to as intention-to-treat (ITT) sample int he HERO study.
Measure: Number; unit: participants
Groups:
- mDOT: mDOT was delivered at both settings and considered a modified version of DOT as not all doses were directly observed
- Patient Navigation: The PN model was developed by the New York City Department of Health and Mental Hygiene. PNs had four roles: (1) coordinating HCV treatment, (2) health education and promotion, (3) assisting participants to overcome personal and structural barriers, and (4) providing psychosocial and adherence support.
Arm/Group | mDOT | Patient Navigation
Number analyzed (Participants) | 376 | 379
participants | 226 | 236

2. Secondary Outcome: HCV DAA Treatment Initiation
Description: (Yes/No). Subject who receive at least one dose of HCV medication (sofosbuvir + velpatasvir) will be considered to have initiated HCV treatment. Those who do not receive one dose within 12 weeks of study enrollment will have been considered not to have initiated HCV treatment.
Time Frame: Up to 12 weeks after study enrollment
Population: ITT sample, that is, all of the participants who were randomized.
Measure: Number; unit: Number of patients who initiated treatme
Arm/Group | mDOT | Patient Navigation
Number analyzed (Participants) | 376 | 379
Number of patients who initiated treatme | 306 | 317

3. Secondary Outcome: Adherence (by Electronic Monitors)
Description: Electronic blister pack data were used to estimate daily adherence, calculated as a binary measure indicating whether one or more doses was taken per day. Weekly adherence levels were then computed in terms of percentages, that is, the number of adherent days out of 7 days for each participant.
Time Frame: During 12 weeks of treatment
Population: mITtT
Measure: Mean (95% Confidence Interval); unit: Percent Adherence
Arm/Group | mDOT | Patient Navigation
Number analyzed (Participants) | 306 | 317
Percent Adherence | 78 [74.8 to 81.4] | 73.4 [70.1 to 76.6]

4. Secondary Outcome: HCV DAA Treatment Completion
Description: (Yes/No) Treatment completion was declared if there were ≥84 days between the treatment initiation and completion.
Time Frame: After 12 weeks of treatment
Population: The number of participants analyzed refer to the number of randomized participants, i.e., the intention-to-treat sample
Measure: Number; unit: # of patients who completed treatment
Arm/Group | mDOT | Patient Navigation
Number analyzed (Participants) | 376 | 379
# of patients who completed treatment | 251 | 264

5. Secondary Outcome: Resistance (to NS5A)
Description: NS5A resistance by Monogram assays.
Time Frame: At weeks 12 or 24
Reporting Status: Not Posted

6. Secondary Outcome: Resistance (to NS5B)
Description: NS5B resistance by Monogram assays
Time Frame: At weeks 12 or 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from baseline to the last visit week, which was 168 weeks after baseline. Therefore, the time frame for the adverse event data collections was 168 weeks, that is slightly longer than 3 years.
Description: An adverse event will be considered serious when the outcome is:
  * Death
  * Life-threatening
  * Hospitalization (initial or prolonged)
  * Disability or permanent damage
  * Congenital Anomaly/Birth Defect
  * Required intervention to prevent permanent impairment or damage (devices)
  * Other serious important medical event
Groups:
- Patient Navigation: The study will follow a PN model (Check Hep C) developed by NYCDOH in collaboration with Montefiore and the community. HCV PNs will provide the following interventions to those randomized to the PN arm: coordination of HCV treatment; health promotion; assisting patients to overcome barriers; and psychosocial support.
  Health Promotion Sessions: PNs will deliver 4 standardized health promotion sessions to all patients either individually or within a group.
Arm/Group | Modified Directly Observed Therapy | Patient Navigation
All-Cause Mortality (participants affected / at risk) | 18/376 | 18/379
Serious Adverse Events (participants affected / at risk) | 6/376 | 11/379
Other Adverse Events (participants affected / at risk) | 3/376 | 2/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Directly Observed Therapy (N=376) | Patient Navigation (N=379)
Hospitalized for kidney stones (Renal and urinary disorders) | 0 | 1
Laceration of right thigh (Injury, poisoning and procedural complications) | 1 | 0
Laryngectomy (Surgical and medical procedures) | 1 | 0
Non-fatal heroin overdose (Injury, poisoning and procedural complications) | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Staph Infection (Skin and subcutaneous tissue disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 5
stab wound - lungs punctured (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Directly Observed Therapy (N=376) | Patient Navigation (N=379)
Tinea cruris (Skin and subcutaneous tissue disorders) | 1 | 0
Itching, crawling skin (Skin and subcutaneous tissue disorders) | 1 | 0
suicidality/psychiatric distress protocol used (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Leg cramps, abdominal discomfort (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT02824640/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT02824640/SAP_001.pdf